CLINICAL TRIAL: NCT02373267
Title: Screening of TMA Patients for ADAMTS13 Activity and the Description of Systematic Organ Damage and/or Organ Failure in Different Entities of Thrombotic Microangiopathies (TMA)
Brief Title: Screening of TMA Patients für ADAMTS13 Activity (Adamscreen)
Acronym: Adamscreen
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. med. Brigitte Schneider, physician, University of Cologne
Other Study IDs: 41-14
Record Dates: First submitted 2015-01-24; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Thrombotic Microangiopathies
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * 2x 5 ml citrate blood
  * 2x 3 ml EDTA blood
  * 1x 5 ml lithium heparin blood
  * 1x 5 ml serum blood
  * 1x 3 ml stool
  * 1x 9 ml urine
  * 1x blood smear
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Technozyme — determination of ADAMTS13 activity

SUMMARY:
Screening of TMA patients for ADAMTS13 activity and the description of systemic organ damage and/or organ failure in different entities of thrombotic microangiopathies (TMA)

DETAILED DESCRIPTION:
This is a prospective diagnostic analysis enrolling 100 patients with clinically suspected thrombotic microangiopathy (TMA) on the basis of laboratory findings such as thrombocytopenia, Coombs negative haemolytic anemia with increased LDH and increased schistozytes. As a first step of differential diagnosis, patients are classified by determining ADAMTS13 activity and antigen concentration and also analyzing for Shigatoxin and Shigatoxin producing bacteria respectively. Primary objective is to determine the relative incidences of the three major entities i.e. aHUS, STEC-HUS and TTP considering distribution of age and gender as well. Mean value of ADAMTS13 activity and antigen measured at date of first diagnosis is considered to line out a threshold value for ADAMTS13 activity pronouncing clinical apparent TMA. Furthermore the present study intends to characterize clinical presentation, clinical course and outcome of different TMA forms particularly with regard to treatment procedures. Monitoring of how ADAMTS13 activity and antigen changes in the course of the disease and in response to treatment is of particular concern for this study. Family history and special clinical conditions should be noted identifying potential genetic predisposition and definite clinical triggers leading to disease manifestation.

ELIGIBILITY:
Inclusion Criteria:

-Patients with first history of TMA as patients with recurrent TMA or TMA in complete or partial remission are eligible for analysis

Exclusion Criteria:

-Patients who received plasma intervention more than 3 weeks prior to screening must be excluded from the observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with a constellation of thrombocytopenia, Coombs negative hemolytic anaemia and clinical signs of ischaemic end organ damage or abdominal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
relative incidences of different entities of TMA | at baseline

SECONDARY OUTCOMES:
Mean value of ADAMTS13 activity and antigen measured at date of first diagnosis. | at baseline

OTHER OUTCOMES:
clinical presentation, clinical course and outcome of different TMA forms particularly with regard to treatment procedures. Monitoring of how ADAMTS13 activity and antigen changes in the course of the disease and in response to treatme | at baseline and in course